CLINICAL TRIAL: NCT04306380
Title: Transoral Incisionless Fundoplication Database Repository (TIF)
Acronym: TIF
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Associate Professor of Medicine, Indiana University
Other Study IDs: 2001738876
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention, database study — data collection from EMR for database

SUMMARY:
Collect data on individuals who have a transoral incisionless fundoplication (TIF) performed by physicians at Indiana University for the treatment of gastroesophageal reflux disease.

DETAILED DESCRIPTION:
Collect patient information related to transoral incisionless fundoplication (TIF) done for gastroesophageal reflux disease. The database information with be used for research to assess trends improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Having a TIF procedure completed at Indiana University Health, University Hospital

Exclusion Criteria:

* under 13 years of age

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Able to give written informed consent and having a TIF procedure for GERD at Indiana University, IU Health university Hospital. Those participants between the age of 13-18 will sign an assent while the parent or guardian will sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
GERD-Health Related Quality of Life Questionnaire (GERD_HRQL) | baseline; 6,12,24 and 60 months
  Change in score for questionnaire related to quality of life with GERD
RESQ-7 questionnaire | baseline; 6,12,24 & 60 months
  Change in score for questionnaire related to symptoms of GERD

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No